CLINICAL TRIAL: NCT02308501
Title: A Single-Center Evaluation of the Anti-Inflammatory Effects of Lastacaft as Measured by In-Vivo Confocal Microscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-100-0012
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-11

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — alcaftadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lastacaft ® (Active Comparator): One drop Lastacaft ® in right eye or left eye based on randomization list once on Day 1 and once on Day 2
  Interventions: Drug: Lastacaft ®
- Tears Naturale ® (Placebo Comparator): One drop Tears Naturale ® in right eye or left eye based on randomization list once on Day 1 and once on Day 2
  Interventions: Drug: Tears Naturale ® (Placebo)

INTERVENTIONS:
Drug: Lastacaft ®
  Arms: Lastacaft ®
Drug: Tears Naturale ® (Placebo)
  Arms: Tears Naturale ®

SUMMARY:
A Single-Center Evaluation of the Anti-Inflammatory Effects of Lastacaft ® as Measured by In-Vivo Confocal Microscopy

ELIGIBILITY:
Inclusion Criteria:

* Have a positive history of ocular allergies and a positive skin test to protocol defined allergens
* Have a positive CAC reaction at Visit 1
* Have a positive conjunctival inflammation score at Visit 1

Exclusion Criteria:

* May not use disallowed medications in specified washout period
* May not have an ocular or system disease the investigator feels with impact subject safety or trial parameters
* May not have active ocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one site in the US.
Pre-assignment Details: Twenty-five participants enrolled and completed the study. Participant flow and baseline characteristics are presented for the 25 subjects (50 participant eyes) that met all inclusion criteria, none of the exclusion criteria and were randomized to receive Lastacaft ® in one eye (25 participant eyes) and Tears Naturale ® (25 participant eyes) in the other based on the randomization list.
Units Other Than Participants: eyes
Groups:
- Lastacaft ®: One drop Lastacaft ® in right eye or left eye based on randomization list once on Day 1 and once on Day 2.
  If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
- Tears Naturale ® (Placebo): One drop Tears Naturale® (Placebo) in right eye or left eye based on randomization list once on Day 1 and once on Day 2. If the right eye was selected for Tears Naturale® (Placebo) at Day 1, the right eye also received Tears Naturale® (Placebo) at Day 2 as dosing did not change between days.
Period: Overall Study
Arm/Group | Lastacaft ® | Tears Naturale ® (Placebo)
Started | 25; 25 eyes (25 participants received one drop of Lastacaft in one eye and Tears Naturale in the other eye.) | 25; 25 eyes
Randomized Participant Eyes | 25; 25 eyes | 25; 25 eyes
Completed | 25; 25 eyes | 25; 25 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: A total of 25 participants enrolled in the study. Since each subject had 1 Lastacaft ® eye and 1 Tears Naturale® eye, the baseline analysis is based on the number of eyes in each arm.
Units Other Than Participants: Eyes
Groups:
- Lastacaft ® Eyes: One drop Lastacaft ® in right eye or left eye based on randomization list once on Day 1 and once on Day 2.
  If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
- Tears Naturale® Eyes: One drop Tears Naturale® (Placebo) in right eye or left eye based on randomization list once on Day 1 and once on Day 2.
  If the right eye was selected for Tears Naturale® (Placebo) at Day 1, the right eye also received Tears Naturale® (Placebo) at Day 2 as dosing did not change between days
- Total: Total of all reporting groups
Arm/Group | Lastacaft ® Eyes | Tears Naturale® Eyes | Total
Number analyzed (Participants) | 25 | 25 | 25
Number analyzed (Eyes) | 25 | 25 | 50
Age, Categorical [Count of Units; unit: Eyes]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 9 | 9 | 18
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: Eyes]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Inflammation at 1 Hour (+30 Minutes) Post CAC on Day 1
Description: Conjunctival Inflammation was assessed by a trained technician post-conjunctival allergen challenge (CAC) on a 0 to 4 scale (0 = best [least inflammation] and 4 = worst [most inflammation]).
  The Conjunctival Inflammation was averaged across all Lastacaft-treated eyes to create the average Lastacaft eye Conjunctival Inflammation score, and the Conjunctival Inflammation score was averaged across all Tears Naturale-treated eyes to create the average Tears Naturale eye Conjunctival Inflammation score.
Time Frame: 1 hour (+30 minutes) post CAC on Day 1
Population: All Randomized Participants Population - All participants who received study treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Lastacaft®: Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of the other treatment in the left eye once on Day 1 based on the randomization list. (participants that received Lastacaft ® in one eye received Tears Naturale® in the other eye at the same time). If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
- Tears Naturale ® (Placebo): Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of the other treatment in the left eye once on Day 1 based on the randomization list. (participants that received Tears Naturale ® in one eye received Lastacaft® in the other eye at the same time). If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
Arm/Group | Lastacaft® | Tears Naturale ® (Placebo)
Number analyzed (Participants) | 25 | 25
Number analyzed (Eyes) | 25 | 25
units on a scale | 3.12 (0.79) | 3.02 (0.80)

2. Primary Outcome: Conjunctival Inflammation 1 Hour (+30 Minutes) Post CAC on Day 2
Description: as for outcome 1
Time Frame: 1 hour (+30 minutes) post CAC on Day 2
Population: All Randomized Participants Population - All participants who received study treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Lastacaft®: Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of the other treatment in the left eye once on Day 2 based on the randomization list. (participants that received Lastacaft ® in one eye received Tears Naturale® in the other eye at the same time). If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
- Tears Naturale ® (Placebo): Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of the other treatment in the left eye once on Day 2 based on the randomization list. (participants that received Tears Naturale ® in one eye received Lastacaft® in the other eye at the same time). If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
Arm/Group | Lastacaft® | Tears Naturale ® (Placebo)
Number analyzed (Participants) | 25 | 25
Number analyzed (Eyes) | 25 | 25
units on a scale | 2.44 (0.97) | 2.90 (0.96)

3. Secondary Outcome: Ocular Itching on Day 1 (15 Minutes Post-study Medication Instillation)
Description: CAC was performed 15 minutes after study medication instillation. Ocular Itching was assessed by the patient on a 0-4 scale (0 = best [no itching] to 4 = worst [severe itching]). The ocular itching score was averaged across all Lastacaft-treated eyes to create the average Lastacaft eye ocular itching score, and the ocular itching score was averaged across all Tears Naturale-treated eyes to create the average Tears Naturale eye ocular itching score.
Time Frame: 15 minutes post-study medication instillation
Population: All Randomized Participants Population - All participants who received study treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Tears Naturale ® (Placebo): Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of the other treatment in the left eye once on Day 1 based on the randomization list. (participants that received Tears Naturale ® in one eye received Lastacaft ® in the other eye at the same time).If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
Arm/Group | Lastacaft® | Tears Naturale ® (Placebo)
Number analyzed (Participants) | 25 | 25
Number analyzed (Eyes) | 25 | 25
units on a scale
  3 minutes post-CAC | 0.72 (0.91) | 2.19 (0.93)
  5 minutes post-CAC | 0.88 (0.92) | 2.41 (0.86)
  7 minutes post-CAC | 0.91 (0.93) | 2.38 (0.90)

4. Secondary Outcome: Ocular Itching on Day 2 (15 Minutes Post-study Medication Instillation)
Description: as for outcome 3
Time Frame: 15 minutes post-study medication instillation
Population: All Randomized Participants Population - All participants who received study treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Tears Naturale® (Placebo): Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of the other treatment in the left eye once on Day 1 based on the randomization list. (participants that received Tears Naturale ® in one eye received Lastacaft® in the other eye at the same time). If the right eye was selected for Lastacaft ® at Day 1, the right eye also received Lastacaft ® at Day 2 as dosing did not change between days.
Arm/Group | Lastacaft® | Tears Naturale® (Placebo)
Number analyzed (Participants) | 25 | 25
Number analyzed (Eyes) | 25 | 25
units on a scale
  3 minutes post-CAC | 0.84 (0.89) | 2.00 (1.02)
  5 minutes post-CAC | 1.16 (0.87) | 2.22 (0.71)
  7 minutes post-CAC | 1.19 (0.85) | 2.22 (0.71)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 5 days. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited, or observed.
Groups:
- Lastacaft®: Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of Lastacaft® or Tears Naturale ® (Placebo) in left eye based on the randomization list. (participants that received Lastacaft ® in one eye received Tears Naturale® in the other eye at the same time)
- Tears Naturale ® (Placebo): Participants received one drop of Lastacaft® or Tears Naturale ® (Placebo) in right eye and one drop of Lastacaft® or Tears Naturale ® (Placebo) in left eye based on the randomization list. (participants that received Tears Naturale ® in one eye received Lastacaft ® in the other eye at the same time)
Arm/Group | Lastacaft® | Tears Naturale ® (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lastacaft® (N=25) | Tears Naturale ® (Placebo) (N=25)
filmy sensation (Eye disorders) | 1 (1) | 1 (1)
blurred vision (Eye disorders) | 1 (1) | 1 (1)
decreased visual acuity (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes